CLINICAL TRIAL: NCT05979207
Title: An Open Label Phase 1b Study to Characterise the Pharmacokinetic/Pharmacodynamic Relationship and Safety of MMV367 in Healthy Adult Participants Experimentally Infected With Blood Stage Plasmodium Falciparum
Brief Title: Phase 1b MMV367 PK/PD and Safety in Healthy Adult Volunteers Experimentally Infected With Blood Stage P. Falciparum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: GlaxoSmithKline (Industry); Southern Star Research (Industry); ICON plc (Industry); QIMR Berghofer Medical Research Institute (Other); Queensland Paediatric Infectious Diseases (QPID) laboratory (Unknown); Swiss BioQuant (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MMV_MMV367_22_01
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Infections; Vector Borne Diseases; Systemic Inflammatory Response Syndrome; Inflammation; Pathologic Processes; Malaria; Malaria,Falciparum; Parasitemia; Parasitic Diseases; Protozoan Infections; Antimalarials; Anti-Infective Agents
Keywords: Malaria; Parasitaemia; Malaria Recrudescence; Malaria, Falciparum
MeSH Terms: conditions — Infections; Vector Borne Diseases; Systemic Inflammatory Response Syndrome; Inflammation; Pathologic Processes; Malaria; Malaria, Falciparum; Parasitemia; Parasitic Diseases; Protozoan Infections

STUDY DESIGN:
Intervention Model Description: MMV367 will be administered as a single oral dose, with different doses to be tested across and within cohorts. The highest dose of MMV367 administered in this study will be no more than 1500 mg, to determine the maximum parasite killing rate of MMV367. Doses to be tested in Cohort 1 will be 20mg, 90mg and 1500mg. Parasite regrowth following initial parasite clearance is required to effectively characterise PK/PD parameters such as the half maximum effective concentration of MMV367.The Safety Data Review Team will review all safety, PK, and PD data. Doses to be tested in Cohort 2 will be informed by the results obtained in Cohort 1, and will be selected to refine the PK/PD parameter estimates. The SDRT will meet following the completion of Cohort 2 to review all safety, PK, and PD data. If the SDRT deems sufficient data has been obtained to achieve the primary endpoint, a third cohort of participants will not be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- MMV367 3mg (Experimental): IBSM challenge and MMV367
  Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. on Day 0 participants will be inoculated intravenously with approximately 2,800 viable P. falciparum-infected erythrocytes.
  Day 8 participants will be dosed with MMV367 when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL.
  Different doses of MMV367 will be administered across and within cohorts in order to effectively characterise the PK/PD relationship.
  Regular safety assessments will be performed and blood will be collected to monitor parasite clearance and MMV367 concentration.
  Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 24, or earlier.
  Interventions: Drug: MMV367 3mg; Other: P. falciparum IBSM infection
- MMV367 5mg (Experimental): IBSM challenge and MMV367
  Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. on Day 0 participants will be inoculated intravenously with approximately 2,800 viable P. falciparum-infected erythrocytes.
  Day 8 participants will be dosed with MMV367 when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL.
  Different doses of MMV367 will be administered across and within cohorts in order to effectively characterise the PK/PD relationship.
  Regular safety assessments will be performed and blood will be collected to monitor parasite clearance and MMV367 concentration.
  Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 24, or earlier.
  Interventions: Other: P. falciparum IBSM infection; Drug: MMV367 5mg
- MMV367 10mg (Experimental): IBSM challenge and MMV367
  Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. on Day 0 participants will be inoculated intravenously with approximately 2,800 viable P. falciparum-infected erythrocytes.
  Day 8 participants will be dosed with MMV367 when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL.
  Different doses of MMV367 will be administered across and within cohorts in order to effectively characterise the PK/PD relationship.
  Regular safety assessments will be performed and blood will be collected to monitor parasite clearance and MMV367 concentration.
  Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 24, or earlier.
  Interventions: Other: P. falciparum IBSM infection; Drug: MMV367 10mg
- MMV367 20mg (Experimental): IBSM challenge and MMV367
  Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. on Day 0 participants will be inoculated intravenously with approximately 2,800 viable P. falciparum-infected erythrocytes.
  Day 8 participants will be dosed with MMV367 when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL.
  Different doses of MMV367 will be administered across and within cohorts in order to effectively characterise the PK/PD relationship.
  Regular safety assessments will be performed and blood will be collected to monitor parasite clearance and MMV367 concentration.
  Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 24, or earlier.
  Interventions: Other: P. falciparum IBSM infection; Drug: MMV367 20mg
- MMV367 90mg (Experimental): IBSM challenge and MMV367
  Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. on Day 0 participants will be inoculated intravenously with approximately 2,800 viable P. falciparum-infected erythrocytes.
  Day 8 participants will be dosed with MMV367 when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL.
  Different doses of MMV367 will be administered across and within cohorts in order to effectively characterise the PK/PD relationship.
  Regular safety assessments will be performed and blood will be collected to monitor parasite clearance and MMV367 concentration.
  Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 24, or earlier.
  Interventions: Other: P. falciparum IBSM infection; Drug: MMV367 90mg
- MMV367 1500mg (Experimental): IBSM challenge and MMV367
  Up to 18 healthy, malaria naïve adult participants are planned to be enrolled into this study, in cohorts of up to six participants each. on Day 0 participants will be inoculated intravenously with approximately 2,800 viable P. falciparum-infected erythrocytes.
  Day 8 participants will be dosed with MMV367 when parasitaemia for the majority of participants is expected to be above 5,000 parasites/mL.
  Different doses of MMV367 will be administered across and within cohorts in order to effectively characterise the PK/PD relationship.
  Regular safety assessments will be performed and blood will be collected to monitor parasite clearance and MMV367 concentration.
  Participants will receive compulsory antimalarial rescue treatment with Riamet® (artemether/lumefantrine) on Day 24, or earlier.
  Interventions: Other: P. falciparum IBSM infection; Drug: MMV367 1500mg

INTERVENTIONS:
Drug: MMV367 3mg — Single dose
  Arms: MMV367 3mg
Other: P. falciparum IBSM infection — Induced Blood Stage Malaria from infected erythrocytes.
Drug: MMV367 5mg — Single dose
  Arms: MMV367 5mg
Drug: MMV367 10mg — Single dose
  Arms: MMV367 10mg
Drug: MMV367 20mg — Single dose
  Arms: MMV367 20mg
Drug: MMV367 90mg — Single dose
  Arms: MMV367 90mg
Drug: MMV367 1500mg — Single dose
  Arms: MMV367 1500mg

SUMMARY:
This is an open-label, adaptive study using the P. falciparum induced blood stage malaria (IBSM) model to characterise the pharmacokinetic/pharmacodynamic (PK/PD) profile and safety of MMV367 (the IMP). Up to 18 participants will be enrolled in cohorts of up to 6 participants each. The study will proceed as follows for all participants:

* Screening period of up to 28 days to recruit healthy adult participants.
* Day 0: Intravenous inoculation with approximately 2,800 viable P. falciparum-infected red blood cells.
* Days 1-3: Daily follow up via phone call or text message.
* Days 4-7: Daily site visits for clinical evaluation and blood sampling to monitor malaria parasite numbers via quantitative polymerase chain reaction (qPCR).
* Day 7 PM: Start of confinement within the clinical trial unit.
* Day 8: Administration of a single oral dose of the IMP (MMV367). Different doses of MMV367 will be administered across and within cohorts in order to effectively characterise the PK/PD relationship.
* Days 8-11: Regular clinical evaluation and blood sampling while confined to monitor malaria parasite numbers and measure MMV367 plasma concentration.
* Day 11 AM: End of confinement within clinical trial unit.
* Days 12-23: Outpatient follow-up for clinical evaluation and blood sampling.
* Day 24: Initiation of compulsory definitive antimalarial treatment with Riamet® (artemether/lumefantrine) and/or other registered antimalarials if required. Treatment will be initiated earlier than Day 24 in the event of:
* Insufficient parasite clearance following IMP dosing
* Parasite regrowth following IMP dosing Characterising the pharmacokinetic/pharmacodynamic relationship of MMV367
* Participant discontinuation/withdrawal,
* Investigator's discretion in the interest of participant safety.
* Day 27: End of study visit for final clinical evaluation and to ensure complete clearance of malaria parasites.

DETAILED DESCRIPTION:
This is an open-label, adaptive study using the P. falciparum induced blood stage malaria (IBSM) model to characterise the pharmacokinetic/pharmacodynamic (PK/PD) profile and safety of MMV367 (the IMP). Up to 18 participants will be enrolled in cohorts of up to 6 participants each. The study will proceed as follows for all participants:

* Screening period of up to 28 days to recruit healthy adult participants.
* Day 0: Intravenous inoculation with approximately 2,800 viable P. falciparum-infected erythrocytes.
* Days 1-3: Daily follow up via phone call or text message.
* Days 4-7: Daily site visits for clinical evaluation and blood sampling to monitor malaria parasitaemia via quantitative polymerase chain reaction (qPCR).
* Day 7 PM: Start of confinement within the clinical trial unit.
* Day 8: Administration of a single oral dose of the IMP (MMV367). Different doses of MMV367 will be administered across and within cohorts in order to effectively characterise the PK/PD relationship.
* Days 8-11: Regular clinical evaluation and blood sampling while confined to monitor malaria parasitaemia and measure MMV367 plasma concentration.
* Day 11 AM: End of confinement within clinical trial unit.
* Days 12-23: Outpatient follow-up for clinical evaluation and blood sampling.
* Day 24: Initiation of compulsory definitive antimalarial treatment with Riamet® (artemether/lumefantrine) and/or other registered antimalarials if required. Treatment will be initiated earlier than Day 24 in the event of:
* Insufficient parasite clearance following IMP dosing (parasitaemia not reduced ≥10-fold by Day 10 compared with peak parasitaemia on Day 8).
* Parasite regrowth following IMP dosing (initial parasite clearance is followed by asexual parasite regrowth above 5000 parasites/mL).

Characterising the pharmacokinetic/pharmacodynamic relationship of MMV367

* Participant discontinuation/withdrawal,
* Investigator's discretion in the interest of participant safety.
* Day 27: End of study visit for final clinical evaluation and to ensure complete clearance of malaria parasitaemia (at least one negative qPCR result required).

ELIGIBILITY:
Inclusion Criteria:

1 Healthy adults aged 18 to 55 years inclusive who will be contactable and available for the duration of the trial and up to two weeks following the EOS visit.

2. Total body weight greater than or equal to 50 kg, and a body mass index (BMI) within the range of 18 to 32 kg/m2 (inclusive). BMI is an estimate of body weight adjusted for height. It is calculated by dividing the weight in kilograms by the square of the height in metres.

3. Completion of the written informed consent process prior to undertaking any trial-related procedure. 4. Must be willing and able to communicate and participate in the whole trial. 5. Agreement to adhere to Lifestyle Considerations (Section 5.3) throughout the trial duration.

6. Must be able to provide contact details of a support person (responsible adult) who is aware of the participant's participation in the study and is available to provide assistance if required (for example with contacting the participant in the event that study staff are unable to, or with transporting the participant to and from the study site if required).

Vital signs and ECG parameters 7. Vital signs at screening (measured after 5 min in the supine position):

* Systolic blood pressure (SBP): 90-140 mmHg,
* Diastolic blood pressure (DBP): 40-90 mmHg,
* Heart rate (HR): 40-100 bpm. Note: Symptomatic postural hypotension will be assessed by measuring SBP and DPB in the standing position (see exclusion criterion 10).

  8. At Screening and pre-inoculation with the malaria challenge agent (Day 0), normal standard mean of triplicate 12-lead electrocardiogram (ECG) parameters after 5 minutes resting in supine position:
* QTcF: ≤450 msec (males) or ≤470 msec (females),
* QRS: 50-120 msec,
* PR interval: ≤ 210 msec,
* Normal ECG tracing unless the Principal Investigator or delegate considers an ECG tracing abnormality to be not clinically relevant.

Contraception 9. Women of childbearing potential (WOCBP) who anticipate being sexually active with a male during the trial must agree to use a highly effective method of birth control (see below) combined with a barrier contraceptive from the screening visit until 34 days after the last dose of MMV367 (covering a full menstrual cycle of 30 days starting after 5 half-lives of last dose of MMV367) and have a negative urine pregnancy test result prior to inoculation with the malaria challenge agent on Day 0.

* Highly effective birth control methods include: combined (oestrogen and progestogen containing) oral/intravaginal/transdermal/implantable hormonal contraception associated with inhibition of ovulation, progestogen-only oral/injectable/implantable hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner, or sexual abstinence or same sex relationship.
* Female participants who are abstinent (from penile-vaginal intercourse) must agree to start a double method if they start a sexual relationship with a male during the study. Female participants must not be planning in vitro fertilisation within the required contraception period.

Women of non-childbearing potential (WONCBP) are defined as:

* Natural (spontaneous) post-menopausal defined as being amenorrhoeic for at least 12 months without an alternative medical cause with a screening follicle stimulating hormone level (FSH) >25 IU/L (or at the local laboratory levels for post-menopause).
* Premenopausal with irreversible surgical sterilization by hysterectomy and/or bilateral oophorectomy or salpingectomy at least 6 months before screening (as determined by participant medical history).

  10. Males who have, or may have, female sexual partners of childbearing potential during the course of the study must agree to use a double method of contraception including condom plus diaphragm, or intrauterine device, or stable oral/transdermal/injectable/implantable hormonal contraceptive by the female partner, from the time of informed consent through to 94 days after MMV367 administration. This has been calculated based on 90 days (one cycle of spermatogenesis) plus 5 half-lives of the IMP (4 days). Abstinent males must agree to start a double method if they begin a sexual relationship with a female during the study and up to 94 days after the last dose of MMV367. Males that are surgically sterile, or who have undergone sterilisation and have had testing to confirm the success of the sterilisation, may also be included and will not be required to use above described methods of contraception.

Exclusion Criteria:

Medical history

1. Known hypersensitivity to artesunate or other artemisinin derivatives, lumefantrine, proguanil/atovaquone, primaquine, or 4-aminoquinolines.
2. Any history of anaphylaxis or other severe allergic reactions, or other food or drug allergy that the Investigator considers may impact on participant safety.
3. History of convulsion (including drug or vaccine-induced episodes). A medical history of febrile convulsion during childhood (< 5 years) is not an exclusion criterion.
4. Presence of current or suspected uncontrolled chronic diseases that may impact participant safety or interpretation of clinical trial results, such as (but not limited to) cardiac or autoimmune disease, diabetes, progressive neurological disease, severe malnutrition, hepatic or renal disease, epilepsy, or asthma.
5. History of malignancy of any organ system (other than localised basal or squamous cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within five years of screening, regardless of whether there is no evidence of local recurrence or metastases.
6. Individuals with history of schizophrenia, bipolar disorder psychoses, attempted or planned suicide, or any other severe (disabling) chronic psychiatric diagnosis including generalised anxiety disorder.
7. History of an episode of depression lasting more than 6 months that required pharmacological therapy and/or psychotherapy within the last 2 years.
8. A score of 20 or more on the Beck Depression Inventory-II (BDI-II) and/or a response of 1, 2 or 3 for item 9 of this inventory (related to suicidal ideation).

   - The BDI-II will be used as a validated tool for the assessment of depression at screening. Participants that meet criterion 8 will be referred to a general practitioner or medical specialist as appropriate. Participants with a BDI-II score of 17 to 19 may be enrolled at the discretion of the Investigator if they do not have a history of the psychiatric conditions mentioned in criterion 6 and their mental state is not considered to pose additional risk to the health of the participant during the trial or to the execution of the trial and interpretation of the data gathered.
9. History of splenectomy.
10. Symptomatic postural hypotension at screening (confirmed on two consecutive readings), irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease of SBP of ≥20 mmHg after 3 min standing and/or a decrease of DBP of ≥10 mmHg after 3 min standing. This 3 min standing period will commence after the volunteer has rested for 5 min in the supine position.
11. Cardiac/QT risk:

    * Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.
    * History of symptomatic cardiac arrhythmias or of clinically relevant bradycardia.
12. Evidence of increased cardiovascular disease risk (defined as >10%, 5-year risk for those greater than 35 years of age, as determined by the Australian Absolute Cardiovascular Disease Risk Calculator [http://www.cvdcheck.org.au/]). Risk factors include sex, age, systolic blood pressure (mm/Hg), smoking status, total and HDL cholesterol (mmol/L), and reported diabetes status.
13. Presence of clinically significant infectious disease or fever (e.g., sublingual temperature ≥38°C) within the five days prior to inoculation.

    Prior medications and treatments
14. Any COVID-19 vaccine within 14 days of malaria inoculation, any other vaccination within 28 days of IMP dosing, and any vaccination planned during the study.
15. Use of prescription drugs (excluding contraceptives), investigational medical products, or nonprescription drugs or herbal supplements, that in the opinion of the investigator may potentially interfere with study interventions, within 14 days or five half-lives (whichever is longer) prior to inoculation. Requirements for concomitant medication use (from inoculation until the end of study) are specified in Section 6.5.
16. Individual who has ever received a blood transfusion. Malaria exposure
17. Any history of malaria or participation in a previous malaria challenge trial or malaria vaccine trial.
18. Must not have had malaria exposure that is considered by the Principal Investigator or their delegate to be significant. This includes but is not limited to: history of having travelled to or lived (>2 weeks) in a malaria-endemic region during the past 12 months or planned travel to a malariaendemic region during the course of the trial; history of having lived for >1 year in a malariaendemic region in the past 10 years; history of having ever lived in a malaria-endemic region for more than 10 years inclusive. For endemic regions see https://malariaatlas.org/explorer/#/, Bali is not considered a malaria-endemic region.

    Alcohol use and smoking
19. History or presence of alcohol abuse (regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type), or drug habituation, or any prior intravenous usage of an illicit substance.
20. Any individual who currently smokes cigarettes on a daily basis (including e-cigarettes, vaping, and other nicotine use).

    Blood donation
21. Blood product donation to any blood bank during the 8 weeks (whole blood) or 4 weeks (plasma and platelets) prior to admission in the clinical unit on Day 8.
22. Individual unwilling to defer blood donations for at least twelve months after the EOS visit.

    Laboratory results
23. Haematology, biochemistry or urinalysis results at screening or at the eligibility visit (Day -1 to Day -3) that are outside of the standard clinically acceptable laboratory ranges (Appendix 12.2) or are considered clinically significant by the Principal Investigator.
24. Positive result for: hepatitis B surface antigen (HBs Ag), anti-hepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab), COVID-19 by PCR at Screening or RAT on Day 0, red blood cell alloantibodies.
25. Positive urine drug test. Any drug listed in the urine drug screen unless there is an explanation acceptable to the Investigator (e.g., the participant has stated in advance that they consumed a prescription or over-the-counter product that contained the detected drug) and the participant has a negative urine drug screen on retest by the pathology laboratory.
26. G6PD deficiency (result below the lower limit of the laboratory reference range for quantitative G6PD test).
27. Positive alcohol breath test.
28. Positive serum pregnancy test at screening or eligibility visit, positive urine pregnancy test on Day 0.

    Other
29. Individual who, in the judgement of the Investigator, is likely to be non-compliant during the trial
30. Individual who is an Investigator, research assistant, pharmacist, trial coordinator, or other staff thereof, directly involved in conducting the trial.
31. Individual without good peripheral venous access.
32. Individual who is breastfeeding or lactating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Bestgen, PhD, Study Director — MMV
Locations (2):
- Australia (2):
  - South Bank, Brisbane, Queensland
  - USC Clinical Trials, Morayfield, Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol allowed for up to 18 participants, that is 3 cohorts of 6 participants, to be enrolled. Between each cohort there was a review of the safety and PK/PD modelling data, before progressing to the next cohort. The review of safety and PK/PD data after cohort 2 determined there was sufficient data to meet the study objective and a third cohort was not required.
Groups:
- Cohort 1: MMV367 20mg: IBSM challenge and MMV367
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
  MMV367 20mg: Single dose
- Cohort 1: MMV367 90mg: IBSM challenge and MMV367
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
  MMV367 90mg: Single dose
- Cohort 1: MMV367 1500mg: IBSM challenge and MMV367
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
  MMV367 1500mg: Single dose
- Cohort 2: MMV367 3mg: IBSM challenge and MMV367
  MMV367 3mg: Single dose
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
- Cohort 2: MMV367 5mg: IBSM challenge and MMV367
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
  MMV367 5mg: Single dose
- Cohort 2: MMV367 10mg: IBSM challenge and MMV367
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
  MMV367 10mg: Single dose
Period: Initial Randomization and PKPD Modelling
Arm/Group | Cohort 1: MMV367 20mg | Cohort 1: MMV367 90mg | Cohort 1: MMV367 1500mg | Cohort 2: MMV367 3mg | Cohort 2: MMV367 5mg | Cohort 2: MMV367 10mg
Started | 3 | 2 | 1 | 0 | 0 | 0
Completed | 3 | 2 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2 Dosing and Modelling
Arm/Group | Cohort 1: MMV367 20mg | Cohort 1: MMV367 90mg | Cohort 1: MMV367 1500mg | Cohort 2: MMV367 3mg | Cohort 2: MMV367 5mg | Cohort 2: MMV367 10mg
Started | 0 | 0 | 0 | 3 | 2 | 1
Completed | 0 | 0 | 0 | 3 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MMV367 3mg: IBSM challenge and MMV367
  MMV367 3mg: Single dose
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
- MMV367 5mg: IBSM challenge and MMV367
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
  MMV367 5mg: Single dose
- MMV367 10mg: IBSM challenge and MMV367
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
  MMV367 10mg: Single dose
- MMV367 20mg: IBSM challenge and MMV367
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
  MMV367 20mg: Single dose
- MMV367 90mg: IBSM challenge and MMV367
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
  MMV367 90mg: Single dose
- MMV367 1500mg: IBSM challenge and MMV367
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
  MMV367 1500mg: Single dose
- Total: Total of all reporting groups
Arm/Group | MMV367 3mg | MMV367 5mg | MMV367 10mg | MMV367 20mg | MMV367 90mg | MMV367 1500mg | Total
Number analyzed (Participants) | 3 | 2 | 1 | 3 | 2 | 1 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.0 (2.00) | 36.5 (17.68) | 33.0 (0) | 23.7 (6.43) | 38.0 (12.73) | 35.0 (0) | 29.0 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 2 | 0 | 1 | 6
  Male | 1 | 1 | 1 | 1 | 2 | 0 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 1 | 3 | 2 | 1 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 1 | 1 | 2 | 2 | 1 | 10
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Multiple | 1 | 1 | 1 | 1 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  Australia | 3 | 2 | 1 | 3 | 2 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Emax
Description: Maximum effect of drug (maximum parasite killing rate). Emax used in the PK/PD model comes from the mean viable parasite elimination half-life of cohort 1 as estimated in the parasite viability report as Emax was not clearly observed in the cohort 2 parasitemia profiles.
Time Frame: Day 8 (IMP dosing) until Day 27 (End of Study)
Population: The model-derived primary outcome Emax is estimated from all reporting groups of cohort 1 and 2.
Measure: Mean (95% Confidence Interval); unit: Maximum clearance rate (1/hour)
Groups:
- IBSM Challenge and MMV367 PK/PD Population Profile: A PK/PD model was built using individual PK parameter estimates of VIS participants as regression parameters to estimate the relationship between MMV367 plasma concentrations, killing and clearance rate of blood stage parasitaemia. A non-linear fixed effects (NLFE) method where population and individual parameters were both treated as fixed effects was used first to test different structural models and obtain initial parameter estimates. (non-linear mixed effects (NLME)was then used with the selected structural model and parameterization as in the NLFE model to estimate the between-subject variability on selected parameters. The MIC, MPC90, and the PRR48max were derived from the final PK/PD model.
Arm/Group | IBSM Challenge and MMV367 PK/PD Population Profile
Number analyzed (Participants) | 6
Maximum clearance rate (1/hour) | 0.35 [0.23 to 0.46]

2. Primary Outcome: EC50
Description: Half Maximal Effective Concentration PK/PD dataset contains the individual information from all arms including date and time of inoculum administration, MMV367 dose; MMV367 plasma PK concentrations; total parasitemia counts by 18S qPCR; gametocytemia counts by pfs25, pfMGET and pfSBP-1 if relevant; and typical covariates such as age, body weight, height, sex and race, to build the model and derive outcome results.
Time Frame: Day 8 (IMP dosing) until Day 27 (End of Study)
Population: Calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan. The PKPD relationship was identified using SysFit as an Emax model with the parameters estimated from the parasitaemia data.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Groups:
- IBSM Challenge and MMV367 PK/PD Population Profile: A PK/PD model was built using individual PK parameter estimates of VIS participants as regression parameters to estimate the relationship between MMV367 plasma concentrations, killing and clearance rate of blood stage parasitaemia. A non-linear fixed effects (NLFE) method where population and individual parameters were both treated as fixed effects was used first to test different structural models and obtain initial parameter estimates. A non-linear mixed effects (NLME) was then used with the selected structural model and parameterization as in the NLFE model to estimate the between-subject variability on selected parameters. The MIC, MPC90, and the PRR48max were derived from the final PK/PD model.
Arm/Group | IBSM Challenge and MMV367 PK/PD Population Profile
Number analyzed (Participants) | 12
ng/mL | 15 [12 to 18]

3. Primary Outcome: MIC
Description: MIC is defined as the concentration when drug killing equals the parasite growth, i.e., the time at which the minimum parasite concentration is observed. Calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan.
Time Frame: Day 8 (IMP dosing) until Day 27 (End of Study)
Population: Calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan.
Measure: Median (95% Confidence Interval); unit: ng/mL
Arm/Group | IBSM Challenge and MMV367 PK/PD Population Profile
Number analyzed (Participants) | 12
ng/mL | 6.3 [5.2 to 7.8]

4. Primary Outcome: MPC90
Description: MPC90 is defined as the concentration at which the clearance effect is at 90% of the maximum. Calculated using the combined data from all doses/arms/groups in both period 1 and 2, as prespecified in section 10 of the Statistical Analysis Plan.
  PK/PD dataset contains the individual information from all arms including date and time of inoculum administration, MMV367 dose; MMV367 plasma PK concentrations; total parasitemia counts by 18S qPCR; gametocytemia counts by pfs25, pfMGET and pfSBP-1 if relevant; and typical covariates such as age, body weight, height, sex and race, to build the model and derive outcome results.
Time Frame: Day 8 (IMP dosing) until Day 27 (End of Study)
Population: as for outcome 3
Measure: Median (Full Range); unit: ng/mL
Arm/Group | IBSM Challenge and MMV367 PK/PD Population Profile
Number analyzed (Participants) | 12
ng/mL | 54 [43 to 68]

5. Primary Outcome: Parasite Killing Achieved Within 48 Hours, PRR48
Description: PRR48 is given as the reduction of values on log10 transformed scale. Only MMV_MMV367_22_01 data was used.
  PRR48 provides an estimate of the efficacy of an anti-malarial treatment. It is the ratio of parasite density over a 48-hour period, estimated using the slope of the optimal fit of the log-linear relationship of parasitemia decay. Optimal fit is derived using geometric mean parasitemia data (i.e. 18S qPCR measuring all blood stage malaria parasites). The optimal fit of the log-linear parasitemia decay by time relationship is determined using left and right censoring to systematically remove potential lag and tail phases of parasitemia decay.
  PRR48 was calculated for each participant using daily PCR data. If the model fit was adequate (overall model p-value<0.001), the slope and corresponding SE from the log-linear regression was used to calculate overall dose-specific PRR48. Participants without adequate model fits were excluded from all dose-specific PRR48 calculations.
Time Frame: Day 8 (IMP dosing) until Day 27 (End of Study)
Population: 2 3mg participants were excluded from the PRR48 calculation and 1 participant was excluded from the 5mg PRR48 calculation due to non-adequate fits.
  Riamet was administered due to parasitaemia and clinical symptoms to participants 108 & 110 [3mg], 107 &112 [5 mg], & 109 [10mg]), parasite regrowth 106 [20mg], or due to positive COVID-19 test (111 [3mg]). 102 & 103 (20mg), 101 & 105 (90mg), & 104 (1500mg) all received definitive antimalarial treatment on Day24 per protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: log[(parasites/mL)/hour]
Groups:
- Cohort 2: MMV367 3mg: IBSM challenge and MMV367
  P. falciparum IBSM infection: Induced Blood Stage Malaria from infected erythrocytes.
  MMV367 3mg: Single dose
Arm/Group | Cohort 1: MMV367 20mg | Cohort 1: MMV367 90mg | Cohort 1: MMV367 1500mg | Cohort 2: MMV367 3mg | Cohort 2: MMV367 5mg | Cohort 2: MMV367 10mg
Number analyzed (Participants) | 3 | 2 | 1 | 1 | 1 | 1
log[(parasites/mL)/hour] | 4.75 [4.29 to 5.20] | 3.64 [3.24 to 4.03] | 4.65 [3.97 to 5.32] | 4.75 [4.17 to 5.34] | 1.81 [1.60 to 2.01] | 2.14 [1.54 to 2.74]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from IMP administration on day 8 until End of Study on day 27.
Description: TEAEs include all AEs reported from the time of IMP dosing to EOS, regardless of relatedness to inoculum or IMP.
Arm/Group | MMV367 3mg | MMV367 5mg | MMV367 10mg | MMV367 20mg | MMV367 90mg | MMV367 1500mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/1 | 0/3 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/1 | 0/3 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/3 | 1/2 | 0/1 | 2/3 | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMV367 3mg (N=3) | MMV367 5mg (N=2) | MMV367 10mg (N=1) | MMV367 20mg (N=3) | MMV367 90mg (N=2) | MMV367 1500mg (N=1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT05979207/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT05979207/SAP_001.pdf
  • Informed Consent Form (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT05979207/ICF_002.pdf